CLINICAL TRIAL: NCT02254993
Title: A Phase 2, Open-Label Study to Evaluate the Safety, Microbiology and Pharmacokinetics of C16G2 Administered in Single or Multiple Oral Gel Doses to Healthy Adult Subjects
Brief Title: Phase 2, Open-Label Study for Safety, Microbiology and PK of Single or Multiple Oral C16G2 Gel Doses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C3J14-201B-00
Record Dates: First submitted 2014-09-24; First posted 2014-10-02 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Arm 1- Part A (Experimental): One 30-minute C16G2 tray gel application (3.2 mg/mL) over the course of five days
  Interventions: Drug: C16G2
- Arm 2 - Part A (Experimental): One 4-hour C16G2 tray gel application (3.2 mg/mL) over the course of five days
  Interventions: Drug: C16G2
- Arm 3- Part A (Experimental): A single 4-hour C16G2 tray gel application (3.2 mg/mL)
  Interventions: Drug: C16G2
- Arm 4- Part A (Experimental): One 4-hour C16G2 tray gel application (1.6 mg/mL) over the course of five days
  Interventions: Drug: C16G2
- Arm 5- Part A (Experimental): One 30-minute C16G2 tray gel application (1.6 mg/mL) over the course of five days
  Interventions: Drug: C16G2
- Arm 6- Part A (Experimental): One 5-minute C16G2 tray gel application (3.2 mg/mL) over the course of five days
  Interventions: Drug: C16G2
- Arm 1 - Part B (Experimental): Four manual brush gel applications on Day 0 followed by twice daily manual brush gel applications (Days 1 through 6); total of 7-day study drug administration, 3.2 mg/mL C16G2 gel concentration.
  Interventions: Drug: C16G2
- Arm 2 - Part B (Experimental): Three manual brush gel applications followed by one tray gel application on Day 0. One manual brush application in the morning and one tray gel application in the evening on Days 1 through 6; total of 7-day study drug administration, 3.2 mg/mL C16G2 gel concentration.
  Interventions: Drug: C16G2
- Arm 3a or 3b or 3c - Part B (Experimental): Based on the microbiology review, one of 3 study arms will be conducted:
  Arm 3a: Four manual brush gel applications on Day 0 followed by twice daily manual brush applications (Days 1 through 6); total of 7-day study drug administration, lower C16G2 concentration of 1.6 mg/mL
  Arm 3b: Three manual brush gel applications followed by one tray gel application on Day 0. One manual brush application in the morning and one tray gel application in the evening on Days 1 through 6; total of 7-day study drug administration, lower C16G2 concentration of 1.6 mg/mL
  Arm 3c: Three daily manual brush and/or tray gel applications for 7 days, lower C16G2 concentration of 1.6 mg/mL
  Interventions: Drug: C16G2
- Arm 4a or 4b - Part B (Experimental): Based on the microbiology review, one of 2 study arms will be conducted:
  Arm 4a: Four manual brush gel applications on Day 0 followed by twice daily manual brush applications (Days 1 through 6); total of 7-day study drug administration, C16G2 concentration of 1.6 mg/mL and lower gel volume
  Arm 4b: Three manual brush gel applications followed by one tray gel application on Day 0. One manual brush application in the morning and one tray gel application in the evening on Days 1 through 6; total of 7-day study drug administration, lower C16G2 concentration of 1.6 mg/mL and lower gel volume
  Interventions: Drug: C16G2
- Arm 5 - Part B (Experimental): Arm 5: Three manual brush gel applications followed by one tray gel application on Day 0, 3.2 mg/mL C16G2 gel concentration.
  Interventions: Drug: C16G2

INTERVENTIONS:
Drug: C16G2 — antimicrobial peptide
  Other Names: C16G2 (1.6 mg/mL); C16G2 (3.2 mg/mL)

SUMMARY:
Part A: Open-label, multiple arm, safety, microbiology and pharmacokinetic (PK) study in healthy adult male and female subjects 18-75 years of age. All subjects will be assessed for safety and microbiology parameters. A subset of subjects will be assessed for pharmacokinetic parameters. No longer enrolling study subjects in Part A.

Part B: Open-label, multiple arm, safety and microbiology study in healthy adult male and female subjects 18-75 years of age. All subjects will be assessed for safety, pharmacokinetic, and microbiology parameters.

DETAILED DESCRIPTION:
Open-label, multiple arm, safety, microbiology and pharmacokinetic (PK) study in healthy adult male and female subjects 18-75 years of age conducted in two parts.

Part A of the study will evaluate up to 6 study arms, depending on the microbiology response evaluated. Before dosing of C16G2, eligible subjects will undergo professional dental prophylaxis on Day 0. Clinic visits for all Study Arms include Visit 1 (Screening/Days -21 to 0), Treatment Visits 2 through 6 (Baseline/Day 0 through Day 4), and follow-up Visits 7 through 11 (Day 5, 8, 12, 19 ± 1 and 33 ± 2).

All subjects will be assessed for safety and microbiology parameters for approximately 5 weeks. A subset of subjects in Study Arms 2 and 4 will be assessed for pharmacokinetic parameters. Part A of the study is no longer enrolling study subjects.

Part B of the study will evaluate up to 5 study arms, depending on the microbiology response evaluated during 2 interim microbiology reviews. Clinic visits for all study arms except Study Arm 5 include Visit 1 (Screening/Days -21 to 0), Visit 2 (Baseline/Day 0), Visits 3 through 17 (Days 1 through 6, morning and evening visits, and Days 7, 10 and 14). All subjects will be assessed for safety and microbiology parameters for approximately 2 weeks. Before dosing of C16G2, eligible subjects will undergo professional dental prophylaxis on Day 0. Study drug will be administered for 7 consecutive days. The Sponsor will perform a microbiology review to evaluate the S. mutans response in Study Arms 1 & 2 and, if applicable, in Study Arms 3a or 3b. In Study Arm 5, subjects will receive multiple C16G2 doses on a single day and will be evaluated for safety, microbiology and pharmacokinetic parameters. Clinic visits for Study Arm 5 will include Visit 1 (Screening/Days -21 to 0), Visit 2 (Baseline/Day 0), Visit 3/Day 1 and Visit 4/Day 6.

ELIGIBILITY:
Inclusion Criteria (Parts A & B):

1. Males and females, 18-75 years of age, inclusive, at the time the Informed Consent Form is signed
2. Female subjects of childbearing potential, defined as not surgically sterile, must agree to use one of the following forms of contraception from screening through the last study visit: hormonal (oral, implant, or injection) begun >30 days prior to screening; barrier (condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD). Acceptable contraceptive options may also include abstinence, monogamous relationship with same sex partner or partner who has had a vasectomy at least six (6) months prior to the screening visit
3. Male subjects only: willing to use contraception or abstain from sexual activity beginning with the first exposure to study drug and continuing until discharged from the study due to completion or Early Termination
4. Healthy, as determined by the Investigator (in consultation with the Medical Monitor, as needed), based on medical and dental history, concurrent illnesses, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (extraoral, head and neck) during Screening
5. Have a minimum of six unrestored bicuspids and molars with ≤50% of molars and bicuspids having restorations, crowns, sealants or are missing
6. Demonstrated ability to expectorate ≥2 mL of stimulated saliva in 5 minutes
7. Have a salivary S. mutans of 2.0 x 10^4 CFUs/mL or greater (Part A) or 1.0 x 10^5 colony forming unit (CFU)/mL or greater (Part B) at Screening using mitis salivarius-bacitracin (MSB) agar plating
8. Willing to refrain from using non-study dentifrice and other non-study oral care products during the study
9. Willing to postpone elective dental procedures (e.g., dental cleanings) between Screening and final post-treatment visit (End of Study or Early Termination)
10. Able to understand and sign the Informed Consent Form prior to initiation of study procedures
11. Able to communicate with the Investigator/study site personnel, understand and comply with the study requirements, and willing to return for protocol-specified visits at the appointed times

Exclusion Criteria (Parts A & B):

1. Advanced periodontal disease
2. Active caries lesion(s) within 30 days prior to study drug administration (confirmed by dental examination and standard radiographs)
3. Medical condition (e.g., artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
4. Pathologic lesions of the oral cavity (suspicious or confirmed)
5. Full or partial dentures, or orthodontic appliances, e.g., night guards, permanent retainers
6. Use of systemic antibiotics, topical oral antibiotics, or use of other drugs, which in the opinion of the Investigator could influence the study outcome, within 30 days prior to Screening
7. Medical history indicating the woman is pregnant, breastfeeding/ lactating or she has a positive urine pregnancy test
8. Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to study drug administration (depending on the specifics, participation in an observational study is not necessarily excluded)
9. Prior participation in a C16G2 clinical trial and known to have received C16G2 active gel or mouth rinse (Note: placebo subjects are not excluded)
10. Presence of any condition or concurrent illness, which in the opinion of the Investigator, would compromise normal immune function (e.g., diabetes, rheumatoid arthritis, lupus, liver disease, organ transplant, etc.), interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of single and multiple C16G2 Gel administrations in healthy adult subjects | All subjects will be monitored for safety for approximately 5 weeks (Visit 2 through Visit 11) in Part A, and for 2 weeks (Visit 2 through 17) in Part B of the study
  Safety will be assessed by comparing the incidence and duration of adverse events, clinically significant changes in vital signs, oral cavity assessments and targeted physical exams in the 6 study arms

SECONDARY OUTCOMES:
To assess antimicrobial activity of C16G2 Gel applications as measured by a reduction in S. mutans in saliva and dental plaque | Visit 2 through Visit 11 (Part A) or Visit 17 (Part B)
  All subjects will be assessed for S. mutans levels for approximately 5 weeks (Part A) or 2 weeks (Part B)
To assess total bacteria in saliva and dental plaque post-study drug administration | Visit 2 through Visit 11 (Part A only)
  All subjects will be assessed for total bacteria levels for approximately 5 weeks (Part A only)
Peak plasma concentration (Cmax) after multiple daily C16G2 Gel administrations | Subjects will be assessed on a single day. PK time points are pre-study drug, during dosing at 5, 30 min, 2 and 4 hrs in Part A and prior to the 1st and 3rd brush, 5 min post 3rd brush, and 15 min and 1.5 hrs after tray
  Five study subjects each in Study Arms 2 and 4 (Part A) and six subjects in Study Arm 5 (Part B). Subjects will be assessed on a single day (Visit 6/Day 4 in Part A and Visit 2/Day 0 in Part B).
Time to peak plasma concentration (Tmax) after multiple daily C16G2 Gel administrations | Subjects will be assessed on a single day. PK time points are pre-study drug, during dosing at 5, 30 min, 2 and 4 hrs in Part A and prior to the 1st and 3rd brush, 5 min post 3rd brush, and 15 min and 1.5 hrs after tray
  Five study subjects each in Study Arms 2 and 4 (Part A) and six subjects in Study Arm 5 (Part B). Subjects will be assessed on a single day (Visit 6/Day 4 in Part A and Visit 2/Day 0 in Part B).
Area under the curve (AUC) after multiple daily C16G2 Gel administrations | Subjects will be assessed on a single day. PK time points are pre-study drug, during dosing at 5, 30 min, 2 and 4 hrs in Part A and prior to the 1st and 3rd brush, 5 min post 3rd brush, and 15 min and 1.5 hrs after tray
  Five study subjects each in Study Arms 2 and 4 (Part A) and six subjects in Study Arm 5 (Part B). Subjects will be assessed on a single day (Visit 6/Day 4 in Part A and Visit 2/Day 0 in Part B).
Volume of distribution (Vd) after multiple daily C16G2 Gel administrations | Subjects will be assessed on a single day. PK time points are pre-study drug, during dosing at 5, 30 min, 2 and 4 hrs in Part A and prior to the 1st and 3rd brush, 5 min post 3rd brush, and 15 min and 1.5 hrs after tray
  Five study subjects each in Study Arms 2 and 4 (Part A) and six subjects in Study Arm 5 (Part B). Subjects will be assessed on a single day (Visit 6/Day 4 in Part A and Visit 2/Day 0 in Part B).
Elimination half life (t 1/2) after multiple daily C16G2 Gel administrations | Subjects will be assessed on a single day. PK time points are pre-study drug, during dosing at 5, 30 min, 2 and 4 hrs in Part A and prior to the 1st and 3rd brush, 5 min post 3rd brush, and 15 min and 1.5 hrs after tray
  Five study subjects each in Study Arms 2 and 4 (Part A) and six subjects in Study Arm 5 (Part B). Subjects will be assessed on a single day (Visit 6/Day 4 in Part A and Visit 2/Day 0 in Part B).
Clearance (Cl) after multiple daily C16G2 Gel administrations | Subjects will be assessed on a single day. PK time points are pre-study drug, during dosing at 5, 30 min, 2 and 4 hrs in Part A and prior to the 1st and 3rd brush, 5 min post 3rd brush, and 15 min and 1.5 hrs after tray
  Five study subjects each in Study Arms 2 and 4 (Part A) and six subjects in Study Arm 5 (Part B). Subjects will be assessed on a single day (Visit 6/Day 4 in Part A and Visit 2/Day 0 in Part B).

CONTACTS AND LOCATIONS:
Overall Officials: Adam D Marberger, DDS, Principal Investigator — Study Center PI; John F Pittaway, DMD, Principal Investigator — Study Center PI
Locations (2):
- United States (2):
  - Plaza West II Dental Group, Kalispell, Montana
  - Jean Brown Research, Salt Lake City, Utah